CLINICAL TRIAL: NCT03199573
Title: Hats on Head Start: A Survey of Sun Protection Behaviors in Head Start and Other Early Childhood Education Programs
Brief Title: Hats on Head Start: A A Survey of Sun Protection Behaviors in Head Start and Other Early Childhood Education Programs
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, Principal Investigator, Northwestern University
Other Study IDs: STU00205541
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Sunburn
Keywords: sunscreen
MeSH Terms: conditions — Sunburn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The proposed study will assess the current sun safety policies and practices in programs for young children and to determine the willingness of stakeholders to incorporate more protective measures.

The primary hypothesis is that children in Head Start programs, daycare programs, elementary schools, or summer camps are exposed to significant UV radiation throughout the day, and are not adequately protected with sunscreen, hats, or sun-protective clothing. The secondary hypothesis is that these programs value sun safety as an important health behavior, but probably do not have the funding avilable to make it a priority.

DETAILED DESCRIPTION:
The study aims are:

1. To assess current exposure to sun and UV in programs of children participating in an early childhood educational program.
2. To assess current policies regarding sun protection and sunscreen use in programs for early childhood education.
3. To assess the current attitudes towards sun safety among caregivers and teachers in programs for early childhood education.
4. To explore association of sun protective behaviors with risk factors such as socioeconomic status, per student classroom budget, program setting (i.e. urban, suburban, or rural), race/ethnicity, size of school program, school budget for supplies, and ages of children enrolled in program.

The sample of stakeholders, who will be surveyed, is consistent with samples used in our prior research. A sample size of 250 phone interviews will be adequate to show trends in sun safety policies among early education programs. Power analysis is based on the use of sun protection, our primary outcome. Our preliminary data show that 15% of schools almost always or always schedule outdoor activities to avoid times when the sun was at peak intensity. The sample size required to sensitively detect a 20% difference in using sun protection between those that comply with recommendations and those that do not is 250 respondents assuming an alpha < 0.05 and power >= 0.8 in a two-tailed test on a two-group sample. This sample size will adequately power the study for detecting 30% difference in sun protection use between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Someone 18 years of age and older, who is a teacher, administrator, aide, or other staff member of a Head Start program, day care program, camp, or elementary school.
* Participants agree to a structured phone interview regarding their program's policies for sun safety, their opinions on certain health behaviors, and the demographics of their student population.
* Participants will be interviewed on the phone and guided through a questionnaire which should take approximately 10 minutes to complete.

Exclusion Criteria:

* Participants who do not know their program's procedures for sun protection will not be able to participate, but may transfer the phone call to another colleague who can answer the questions accurately. Participants without the ability to speak in English will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Teachers, aides, administrators or staff members at Head Start programs, daycares, camps, or schools.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Total daily sun exposure and sunburn of children | 10 minutes
  Total sun exposure per day and number of sunburns sustained at Head Start program, daycare, camp, or school

SECONDARY OUTCOMES:
Sun safety policies | 10 minutes
  presence of policies in place to protect children from UV exposure e.g. designated time to don sun protective clothing, encouraging parents to apply sunscreen before school, send children with sun hats.

OTHER OUTCOMES:
Demographics | 10 minutes
  Demographics of programs contacted e.g. racial breakdown, socioeconomic status of families served, ages of children in program, setting.

CONTACTS AND LOCATIONS:
Overall Officials: June Robinson, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guy GP Jr, Thomas CC, Thompson T, Watson M, Massetti GM, Richardson LC; Centers for Disease Control and Prevention (CDC). Vital signs: melanoma incidence and mortality trends and projections - United States, 1982-2030. MMWR Morb Mortal Wkly Rep. 2015 Jun 5;64(21):591-6. PMID 26042651
- [Background] Rogers HW, Weinstock MA, Feldman SR, Coldiron BM. Incidence Estimate of Nonmelanoma Skin Cancer (Keratinocyte Carcinomas) in the U.S. Population, 2012. JAMA Dermatol. 2015 Oct;151(10):1081-6. doi: 10.1001/jamadermatol.2015.1187. PMID 25928283
- [Background] Gandini S, Sera F, Cattaruzza MS, Pasquini P, Picconi O, Boyle P, Melchi CF. Meta-analysis of risk factors for cutaneous melanoma: II. Sun exposure. Eur J Cancer. 2005 Jan;41(1):45-60. doi: 10.1016/j.ejca.2004.10.016. PMID 15617990
- [Background] Godar DE, Urbach F, Gasparro FP, van der Leun JC. UV doses of young adults. Photochem Photobiol. 2003 Apr;77(4):453-7. doi: 10.1562/0031-8655(2003)0772.0.co;2. PMID 12733658
- [Background] Buller DB, Borland R. Skin cancer prevention for children: a critical review. Health Educ Behav. 1999 Jun;26(3):317-43. doi: 10.1177/109019819902600304. PMID 10349571
- [Background] Buller DB, Geller AC, Cantor M, Buller MK, Rosseel K, Hufford D, Benjes L, Lew RA. Sun protection policies and environmental features in US elementary schools. Arch Dermatol. 2002 Jun;138(6):771-4. doi: 10.1001/archderm.138.6.771. PMID 12056958
- [Background] Shanklin S, Brener ND, Kann L, Griffin-Blake S, Ussery-Hall A, Easton A, Barrett E, Hawkins J, Harris WA, McManu T; Centers for Disease Control and Prevention (CDC). Youth risk behavior surveillance--selected Steps communities, United States, 2007. MMWR Surveill Summ. 2008 Nov 21;57(12):1-27. PMID 19023264
- [Background] Hall HI, Jorgensen CM, McDavid K, Kraft JM, Breslow R. Protection from sun exposure in US white children ages 6 months to 11 years. Public Health Rep. 2001 Jul-Aug;116(4):353-61. doi: 10.1093/phr/116.4.353. PMID 12037264
- [Background] Cokkinides V, Weinstock M, Glanz K, Albano J, Ward E, Thun M. Trends in sunburns, sun protection practices, and attitudes toward sun exposure protection and tanning among US adolescents, 1998-2004. Pediatrics. 2006 Sep;118(3):853-64. doi: 10.1542/peds.2005-3109. PMID 16950974
- [Background] Buller DB, Cokkinides V, Hall HI, Hartman AM, Saraiya M, Miller E, Paddock L, Glanz K. Prevalence of sunburn, sun protection, and indoor tanning behaviors among Americans: review from national surveys and case studies of 3 states. J Am Acad Dermatol. 2011 Nov;65(5 Suppl 1):S114-23. doi: 10.1016/j.jaad.2011.05.033. PMID 22018060
- [Background] Buller DB, Hall JR, Powers PJ, Ellsworth R, Beach BH, Frank CA, Maloy JA, Buller MK. Evaluation of the "Sunny Days, Healthy Ways" sun safety CD-ROM program for children in grades 4 and 5. Cancer Prev Control. 1999 Jun;3(3):188-95. PMID 10474766
- [Background] Buller DB, Taylor AM, Buller MK, Powers PJ, Maloy JA, Beach BH. Evaluation of the Sunny Days, Healthy Ways sun safety curriculum for children in kindergarten through fifth grade. Pediatr Dermatol. 2006 Jul-Aug;23(4):321-9. doi: 10.1111/j.1525-1470.2006.00270.x. PMID 16918625
- [Background] Hewitt M, Denman S, Hayes L, Pearson J, Wallbanks C. Evaluation of 'Sun-safe': a health education resource for primary schools. Health Educ Res. 2001 Oct;16(5):623-33. doi: 10.1093/her/16.5.623. PMID 11675809
- [Background] Giles-Corti B, English DR, Costa C, Milne E, Cross D, Johnston R. Creating SunSmart schools. Health Educ Res. 2004 Feb;19(1):98-109. doi: 10.1093/her/cyg003. PMID 15020549
- [Background] Buller DB, Borland R. Public education projects in skin cancer prevention: child care, school, and college-based. Clin Dermatol. 1998 Jul-Aug;16(4):447-59. doi: 10.1016/s0738-081x(98)00018-2. No abstract available. PMID 9699057
- [Background] Buller DB, Burgoon M, Hall JR, Levine N, Taylor AM, Beach B, Buller MK, Melcher C. Long-term effects of language intensity in preventive messages on planned family solar protection. Health Commun. 2000;12(3):261-75. doi: 10.1207/S15327027HC1203_03. PMID 10938916
- [Background] English DR, Milne E, Jacoby P, Giles-Corti B, Cross D, Johnston R. The effect of a school-based sun protection intervention on the development of melanocytic nevi in children: 6-year follow-up. Cancer Epidemiol Biomarkers Prev. 2005 Apr;14(4):977-80. doi: 10.1158/1055-9965.EPI-04-0531. PMID 15824173
- [Background] Geller AC, Shamban J, O'Riordan DL, Slygh C, Kinney JP, Rosenberg S. Raising sun protection and early detection awareness among Florida high schoolers. Pediatr Dermatol. 2005 Mar-Apr;22(2):112-8. doi: 10.1111/j.1525-1470.2005.22204.x. PMID 15804297
- [Background] Norman GJ, Adams MA, Calfas KJ, Covin J, Sallis JF, Rossi JS, Redding CA, Cella J, Patrick K. A randomized trial of a multicomponent intervention for adolescent sun protection behaviors. Arch Pediatr Adolesc Med. 2007 Feb;161(2):146-52. doi: 10.1001/archpedi.161.2.146. PMID 17283299
- [Background] Buller MK, Kane IL, Martin RC, Giese AJ, Cutter GR, Saba LM, Buller DB. Randomized trial evaluating computer-based sun safety education for children in elementary school. J Cancer Educ. 2008;23(2):74-9. doi: 10.1080/08858190701818267. PMID 18569241
- [Background] Glanz K, Saraiya M, Wechsler H; Centers for Disease Control and Prevention. Guidelines for school programs to prevent skin cancer. MMWR Recomm Rep. 2002 Apr 26;51(RR-4):1-18. PMID 11995901
- [Background] Emmons KM, Colditz GA. Preventing excess sun exposure: it is time for a national policy. J Natl Cancer Inst. 1999 Aug 4;91(15):1269-70. doi: 10.1093/jnci/91.15.1269. No abstract available. PMID 10433608
- [Background] Grunbaum JA, Rutman SJ, Sathrum PR. Faculty and staff health promotion: results from the School Health Policies and Programs Study 2000. J Sch Health. 2001 Sep;71(7):335-9. doi: 10.1111/j.1746-1561.2001.tb03512.x. No abstract available. PMID 11586876
- [Background] Tang KC, Beaglehole R, O'Byrne D. Policy and partnership for health promotion--addressing the determinants of health. Bull World Health Organ. 2005 Dec;83(12):884. Epub 2006 Jan 30. No abstract available. PMID 16462974
- [Background] French SA, Jeffery RW, Story M, Breitlow KK, Baxter JS, Hannan P, Snyder MP. Pricing and promotion effects on low-fat vending snack purchases: the CHIPS Study. Am J Public Health. 2001 Jan;91(1):112-7. doi: 10.2105/ajph.91.1.112. PMID 11189801
- [Background] French SA, Story M, Fulkerson JA. School food policies and practices: a state-wide survey of secondary school principals. J Am Diet Assoc. 2002 Dec;102(12):1785-9. doi: 10.1016/s0002-8223(02)90382-2. PMID 12487541
- [Background] Hinman AR, Orenstein WA, Williamson DE, Darrington D. Childhood immunization: laws that work. J Law Med Ethics. 2002 Fall;30(3 Suppl):122-7. PMID 12508514
- [Background] Glanz K, Lankenau B, Foerster S, Temple S, Mullis R, Schmid T. Environmental and policy approaches to cardiovascular disease prevention through nutrition: opportunities for state and local action. Health Educ Q. 1995 Nov;22(4):512-27. doi: 10.1177/109019819502200408. PMID 8550374
- [Background] Buller DB, Buller MK, Reynolds KD. A survey of sun protection policy and education in secondary schools. J Am Acad Dermatol. 2006 Mar;54(3):427-32. doi: 10.1016/j.jaad.2005.11.1030. Epub 2006 Jan 23. PMID 16488293
- [Background] Everett Jones S, Guy GP Jr. Sun Safety Practices Among Schools in the United States. JAMA Dermatol. 2017 May 1;153(5):391-397. doi: 10.1001/jamadermatol.2016.6274. PMID 28257534